CLINICAL TRIAL: NCT03828968
Title: Chronic Urinary Retention in Elderly Living in Homes for the Aged : Benefits of Bladder Scan Screening
Acronym: RUC EHPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC18_3063_RUC EHPAD
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Urinary Retention
Keywords: urinary retention; chronic disease; aged; homes for the aged
MeSH Terms: conditions — Urinary Retention; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bladder scan (Other): Bladder scan performed on resident in homes for aged
  Interventions: Diagnostic Test: bladder scan

INTERVENTIONS:
Diagnostic Test: bladder scan — Measurement of vesical volume by bladder scan

SUMMARY:
The goal of this cross-sectional, multicentric and descriptive epidemiological study is to assess the prevalence of chronic urinary retention (CUR) in elderly living in residential care for dependent elderly people in order to determine if there is an interest in offering them a bladder scan screening.

DETAILED DESCRIPTION:
The main goal of this study is to assess the prevalence of CUR in elderly living in homes for the aged, the secondary ones are to evaluate the risk factors and complications of CUR.

We will carry out this prevalence study in 5 centres whit a draw of 40 residents per centre. Following an information and a non-opposition of the patients, we will collect datas in their medical file (age, medical history and comorbidities, current treatments, anticholinergic score according to the ADS (Anticholinergic Drug Scale), GIR score according to the AGGIR scale (Autonomie Gérontologique Groupes Iso Ressources), FAC modified score (Functional Ambulation Classification modified), MMSE score (Mini Mental State Examination), communicative capacity, notion of fall and date of last fall, knowledge of urinary incontinence, knowledge of constipation, knowledge of previous urinary screening by bladder scan and previous urological consulting, last urinalysis and its results, last analysis of creatinemia and creatinine clearance according to CKD-EPI) and we will perform up to 3 measurements of vesical volume by bladder scan.

The expected results are a prevalence of CUR between 10 and 20 % among people living in homes for the aged with more urinary tract infections, renal insufficiency and falls in the CUR group showing the interest of screening for CUR by bladder scan in elderly people living in nursing homes according to risk groups based on the risk factors found.

ELIGIBILITY:
Inclusion Criteria:

* Adult people
* Residents in a participating nursing home

Exclusion Criteria:

* Resident with indwelling urinary catheter or regular urinary catheterisation
* Resident or legal representative opposing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Chronic urinary retention | 4 weeks after inclusion
  Chronic urinary retention definition : post-void residual urine > 250 mL twice without any clinical argument for acute urinary retention.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud HONORE, MD, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - EHPAD du Centre Local Hospitalier de Saint-Joseph, Combourg
  - EHPAD du Centre Hospitalier de Fougères, Fougères
  - EHPAD Hôtel-Dieu, Rennes
  - EHPAD de Saint-Brice-en-Coglès, Saint-Brice-en-Coglès
  - EHPAD de Saint-Georges-de-Reintembault, Saint-Georges-de-Reintembault